CLINICAL TRIAL: NCT00289640
Title: A Randomized, Double-Blind, Multi-center, Phase II Fixed Dose Study of Multiple Doses of Ipilimumab (MDX-010) Monotherapy in Patients With Previously Treated Unresectable Stage III or IV Melanoma
Brief Title: Study of Ipilimumab (MDX-010) Monotherapy in Patients With Previously Treated Unresectable Stage III or IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA184-022
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2009-01

CONDITIONS: Melanoma
Keywords: Stage III (unresectable); Stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: ipilimumab (MDX-010, BMS-734016)
- 2 (Experimental)
  Interventions: Drug: Ipilimumab
- 3 (Experimental)
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: ipilimumab (MDX-010, BMS-734016) — IV solution, IV, 0.3mg/kg, Q 3 wks for 12 wks then Q 12 wks, 48+ weeks depending on response.
  Arms: 1
Drug: Ipilimumab — IV solution, IV, 3 mg/kg, Q 3 wks for 12 wks then Q 12 wks, 48+ weeks depending on response.
  Arms: 2
Drug: Ipilimumab — IV solution, IV, 10 mg/kg, Q 3 wks for 12 wks then Q 12 wks, 48+ weeks depending on response.
  Arms: 3

SUMMARY:
The purpose of this clinical research study is to compare the best overall response rate (BORR)(as per modified WHO criteria) in patients with previously treated, therapy-refractory, or -intolerant, Stage III (unresectable) or Stage IV melanoma receiving ipilimumab doses of 0.3, 3, and 10 mg/kg. The safety of this product will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously treated, therapy-refractory or -intolerant, Stage III (unresectable) or Stage IV melanoma

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
estimate BORR in patients with previously treated, therapy-refractory or -intolerant, Stage III (unresectable) or Stage IV melanoma receiving ipilimumab doses of 0.3, 3, and 10 mg/kg.

SECONDARY OUTCOMES:
estimate progression free survival rate at Week 12 assessment and other timepoints
estimate disease control rate at various time points
estimate overall survival
estimate survival rate at one year
evaluate health-related quality of life
obtain pharmacokinetic samples for population PK analysis

CONTACTS AND LOCATIONS:
Locations (58):
- United States (25):
  - Arizona Cancer Center, Tucson, Arizona
  - Wilshire Oncology Medical Group Inc, Laverne, California
  - Scripps Cancer Center, San Diego, California
  - The Angeles Clinic And Research Institution, Santa Monica, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Baptist Cancer Institute, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Md Anderson Cancer Center Orlando, Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Oncology Specialists, Sc, Park Ridge, Illinois
  - American Health Network, Indianapolis, Indiana
  - University Of Louisville, Louisville, Kentucky
  - Harry And Jeanette Weinberg Cancer Inst At Franklin Square, Baltimore, Maryland
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - St Joseph Oncology Inc, Saint Joseph, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - The Christ Hospital Cancer Center Research, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Cancer Centers Of The Carolinas, Greenville, South Carolina
  - Center For Oncology Research & Treatment, P.A., Dallas, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
- Australia (4):
  - Local Institution, Newcastle, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Wodonga, Victoria
- Local Institution, Brussels, Belgium
- Brazil (4):
  - Local Institution, Centro-Porto Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Jaú, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (3):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Kingston, Ontario
- Czechia (2):
  - Local Institution, Olomouc
  - Local Institution, Prague
- France (8):
  - Local Institution, Brest, Cedex
  - Local Institution, Clermont-Ferrand
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Rennes
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (7):
  - Local Institution, Berlin
  - Local Institution, Essen
  - Local Institution, Heidelberg
  - Local Institution, Jena
  - Local Institution, Kiel
  - Local Institution, Mannheim
  - Local Institution, Würzburg
- Local Institution, Pécs, Hungary
- South Africa (3):
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Cape Town, Western Cape

REFERENCES:
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Derived] Wolchok JD, Neyns B, Linette G, Negrier S, Lutzky J, Thomas L, Waterfield W, Schadendorf D, Smylie M, Guthrie T Jr, Grob JJ, Chesney J, Chin K, Chen K, Hoos A, O'Day SJ, Lebbe C. Ipilimumab monotherapy in patients with pretreated advanced melanoma: a randomised, double-blind, multicentre, phase 2, dose-ranging study. Lancet Oncol. 2010 Feb;11(2):155-64. doi: 10.1016/S1470-2045(09)70334-1. Epub 2009 Dec 8. PMID 20004617